CLINICAL TRIAL: NCT00915551
Title: A Multi-center, Randomized, Parallel Group, Double-blind, Vehicle-controlled Study to Evaluate the Efficacy and Safety of PEP005 (Ingenol Mebutate) Gel, 0.015% In Patients With Actinic Keratoses ON the Head (Face or Scalp) (REGION-IIb)
Brief Title: A Multi-Center Study to Evaluate the Efficacy and Safety of PEP005 (Ingenol Mebutate) Gel, When Used to Treat Actinic Keratoses on the Head (Face or Scalp)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEP005-025
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2013-11

CONDITIONS: Actinic Keratosis
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP005 (Ingenol Mebutate) gel (Experimental)
  Interventions: Drug: PEP005 (Ingenol Mebutate) gel, 0.015%
- Vehicle gel (Placebo Comparator)
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: PEP005 (Ingenol Mebutate) gel, 0.015% — once daily for 3 consecutive days
  Arms: PEP005 (Ingenol Mebutate) gel
Drug: Vehicle Gel — once daily for 3 consecutive days
  Arms: Vehicle gel

SUMMARY:
This Phase III study is designed to assess the efficacy and safety of PEP005 Gel, 0.015% when applied to an area of skin containing 4-8 AK lesions on the face or scalp.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and at least 18 years of age
* Female patients must be of either:

  * Non-childbearing potential, post-menopausal
  * Childbearing potential, provided there are negative serum and urine pregnancy test results prior to study treatment, to rule out pregnancy

Exclusion Criteria:

* Cosmetic or therapeutic procedures within 2 weeks and 2cm of the selected treatment area
* Treatment with immunomodulators, or interferon/ interferon inducers or systemic medications that suppress the immune system within 4 weeks
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy: within 8 weeks and 2 cm of the selected treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (19):
  - Burke Pharmaceutical Research, Hot Springs, Arizona
  - Center for Dermatology, Fremont, California
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Laser Skin Surgery Center of Indiana, Carmel, Indiana
  - Deaconess Clinic, Inc, Evansville, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Skin Specialists, PC, Omaha, Nebraska
  - Karl G. Heine Dermatology, Henderson, Nevada
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - Dermatology Associates of Rochester, PC, Rochester, New York
  - Dermatology, Laser Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Oregon Medical Research Center, PC, Portland, Oregon
  - DermResearch, Inc., Austin, Texas
  - Suzanne Bruce and Associates, PA, The Center for Skin Research, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - The Education and Research Foundation, Lynchburg, Virginia
  - Premier Clinical Research, Spokane, Washington
- Australia (2):
  - The Skin Centre, Benowa, Queensland
  - South East Dermatology, Belmont Specialist Centre, Carina Heights, Queensland

REFERENCES:
- [Derived] Lebwohl M, Swanson N, Anderson LL, Melgaard A, Xu Z, Berman B. Ingenol mebutate gel for actinic keratosis. N Engl J Med. 2012 Mar 15;366(11):1010-9. doi: 10.1056/NEJMoa1111170. PMID 22417254
- See also: Food and Drug Authority — http://www.fda.gov
- See also: Therapeutic Goods Administration — http://www.tga.gov.au

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study PEP005-025 was conducted at 21 study centers in the United States (19) and Australia (2). A total of 278 patients were randomized (255 (92%) in the US and 23 (8%) in Australia). Patient screening was started on 05 May 2009. The first patient was randomized on 05 June 2009 and the last patient completed the Day 57 visit on 02 September 2009.
Groups:
- PEP005 (Ingenol Mebutate) Gel, 0.015%: PEP005 (ingenol mebutate) Gel 0.05% once daily for 3 consecutive days
- Vehicle Gel: Vehicle gel once daily for 3 consecutive days
Period: Overall Study
Arm/Group | PEP005 (Ingenol Mebutate) Gel, 0.015% | Vehicle Gel
Started | 142 | 136
Completed | 142 | 135
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEP005 (Ingenol Mebutate) Gel, 0.015% | Vehicle Gel | Total
Number analyzed (Participants) | 142 | 136 | 278
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 63 | 136
  >=65 years | 69 | 73 | 142
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 117 | 112 | 229
Region of Enrollment [Number; unit: participants]
  United States | 131 | 124 | 255
  Australia | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance of Actinic Keratoses (AK) Lesions
Description: Complete clearance of the treatment field
Time Frame: baseline and 57 days
Population: Intention to treat population
Measure: Number; unit: participants
Groups:
- PEP005 (Ingenol Mebutate) Gel, 0.015%: PEP005 (Ingenol Mebutate) gel, 0.015% once daily for 3 consecutive days
Arm/Group | PEP005 (Ingenol Mebutate) Gel, 0.015% | Vehicle Gel
Number analyzed (Participants) | 142 | 136
participants | 67 [upper limit 55.7] | 7 [2.1 to 10.3]
Statistical Analysis 1: Comparison: PEP005 (Ingenol Mebutate) Gel, 0.015% vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Partial Clearance of Actinic Keratoses (AK)
Description: Partial clearance defined as ≥ 75% reduction in the number of AK lesions identified at baseline in the treatment area
Time Frame: baseline and 57 days
Population: Intention to treat population
Measure: Number; unit: participants
Arm/Group | PEP005 (Ingenol Mebutate) Gel, 0.015% | Vehicle Gel
Number analyzed (Participants) | 142 | 136
participants | 96 | 11
Statistical Analysis 1: Comparison: PEP005 (Ingenol Mebutate) Gel, 0.015% vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 57 days
Arm/Group | PEP005 (Ingenol Mebutate) Gel, 0.015% | Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 1/142 | 0/136
Other Adverse Events (participants affected / at risk) | 20/142 | 1/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEP005 (Ingenol Mebutate) Gel, 0.015% (N=142) | Vehicle Gel (N=136)
Hip Arthroplasty (Hip Replacement) (Surgical and medical procedures) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEP005 (Ingenol Mebutate) Gel, 0.015% (N=142) | Vehicle Gel (N=136)
Application site pain (Skin and subcutaneous tissue disorders) | 17 | 1
Application site pruritus (Skin and subcutaneous tissue disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For US sites: The institution and investigator agree not to publish the results of this study without prior written consent of the Sponsor. As used herein, the term "publish" shall include oral presentations,written abstracts, written manuscripts, etc.